CLINICAL TRIAL: NCT00691197
Title: Safety and Acceptability of Using a Rewetting Drop With Contact Lens Wear
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG9689-002
Record Dates: First submitted 2008-03-04; First posted 2008-06-05 (Estimated); Results first posted 2009-12-10 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carboxymethylcellulose sodium and Glycerin (Experimental): Carboxymethylcellulose sodium and Glycerin based rewetting drop
  Interventions: Device: Carboxymethylcellulose sodium and Glycerin
- Carboxymethylcellulose sodium (Active Comparator): Carboxymethylcellulose sodium based rewetting drop
  Interventions: Device: Carboxymethylcellulose sodium

INTERVENTIONS:
Device: Carboxymethylcellulose sodium and Glycerin — Eye drops used at least 4 times per day, 1-2 drops in each eye while wearing contact lenses.
  Other Names: Optive™
  Arms: Carboxymethylcellulose sodium and Glycerin
Device: Carboxymethylcellulose sodium — Eye drops used at least 4 times per day, 1-2 drops in each eye while wearing contact lenses.
  Other Names: Refresh Contacts®
  Arms: Carboxymethylcellulose sodium

SUMMARY:
Testing the Safety and Acceptability of Using a Rewetting Drop with Contact Lenses

ELIGIBILITY:
Inclusion Criteria:

* Adapted contact lens wearer

Exclusion Criteria:

* Monovision lens wearer, ocular or systemic disease, pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Allergan
Locations (1):
- San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboxymethylcellulose Sodium and Glycerin | Carboxymethylcellulose Sodium
Started | 166 | 80
Completed | 155 | 75
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose Sodium and Glycerin | Carboxymethylcellulose Sodium | Total
Number analyzed (Participants) | 166 | 80 | 246
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.6 (11.94) | 36.8 (11.54) | 37.4 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 53 | 175
  Male | 44 | 27 | 71

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity
Description: Percentage of Subjects Tabulated by Changes in Line Number at Day 90 from Baseline; Visual Acuity measured by LogMar reported as Snellen equivalents. Better: an increase of 2 lines or more in at least one eye; No Change: a change less than +/- 2 lines in both eyes; Worse: a decrease of 2 lines or more in at least one eye.
Time Frame: Change from Baseline at Day 90
Population: Completed Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Carboxymethylcellulose Sodium and Glycerin | Carboxymethylcellulose Sodium
Number analyzed (Participants) | 155 | 75
Percentage of Participants
  Better | 0.65 | 1.33
  No Change | 98.06 | 98.67
  Worse | 1.29 | 0

2. Post Hoc Outcome: Patient Acceptability
Description: A questionnaire was administered to all patients to evaluate the acceptability of the Rewetting Drops (RD) with use with Contact Lenses (CL). Table below shows the percentage of participants responding either "Agree" or "Strongly Agree" at day 90. Number of participants answering question is indicated as (number of Test subjects/number of Control subjects)
Time Frame: Day 90
Population: Intent to Treat Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Carboxymethylcellulose Sodium and Glycerin | Carboxymethylcellulose Sodium
Number analyzed (Participants) | 161 | 79
Percentage of Participants
  Liked using the RD (160/78) | 72.5 | 82.1
  RD gave good comfort during day (161/79) | 78.8 | 84.8
  RD on CL gave good initial comfort (161/79) | 49.0 | 54.4
  At day's end,CL felt better after RD use (161/78) | 51.6 | 62.8
  Could wear CL longer when using RD (161/79) | 46.6 | 44.3
  Vision was normal soon after using RD (161/79) | 85.7 | 81.0
  Vision with CL was better after RD use (161/79) | 31.0 | 41.8
  Would likely purchase these RD (161/79) | 50.4 | 68.4
  Eyes felt better after CL removal (161/79) | 38.5 | 43.1

3. Secondary Outcome: Corneal Staining
Description: Corneal staining of greater or equal to grade 2 at day 90. Grading scale: 0 = None Present; 1 = Trace Finding; 2 = Mild Finding; 3 = Moderate Finding; 4 = Severe Finding
Time Frame: Day 90
Population: Completed Population
Measure: Number; unit: Participants
Arm/Group | Carboxymethylcellulose Sodium and Glycerin | Carboxymethylcellulose Sodium
Number analyzed (Participants) | 155 | 75
Participants | 0 | 1

4. Post Hoc Outcome: Patient Preference
Description: Percentage of patients who used pre-study rewetting drops and answered "Agree" or "Strongly Agree" when asked if they preferred the study drops (SD) over their pre-study drops(PSD).
Time Frame: Day 30
Population: Responders Completed Population
Measure: Number; unit: Percentage of participants
Arm/Group | Carboxymethylcellulose Sodium and Glycerin | Carboxymethylcellulose Sodium
Number analyzed (Participants) | 79 | 41
Percentage of participants
  Prefer SD over PSD | 47.2 | 41.5
  SD more comfortable overall than PSD | 53.2 | 34.1

ADVERSE EVENTS:
Arm/Group | Carboxymethylcellulose Sodium and Glycerin | Carboxymethylcellulose Sodium
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/79
Other Adverse Events (participants affected / at risk) | 15/166 | 11/79
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboxymethylcellulose Sodium and Glycerin (N=166) | Carboxymethylcellulose Sodium (N=79)
Asthenopia (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 2 | 2
Eye discharge (Eye disorders) | 3 | 0
Eye irritation (Eye disorders) | 3 | 1
Ocular discomfort (Eye disorders) | 2 | 0
Conjunctival oedema (Eye disorders) | 1 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Episcleritis (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 2
Limbal hyperaemia (Eye disorders) | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 90 days from the time submitted to the sponsor for review.

The sponsor cannot require changes to the communication and cannot extend the embargo.